CLINICAL TRIAL: NCT05964530
Title: Comparing the Oncologic Efficacy of Radical Versus Local Excision for Rectal Cancer With Clinically Complete Remission to Neoadjuvant Chemoradiation Therapy: A Randomized Controlled Clinical Trial
Brief Title: Radical vs Local Excision for Rectal Cancer With Clinically Complete Remission
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202212114RIND
Record Dates: First submitted 2023-07-17; First posted 2023-07-28 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Concomitant chemoradiation therapy; Radical surgery; Local excision
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watch and wait group (Experimental): In this group, the patients with clinically complete response will undergo non-surgical treatment (watch-and-wait group)
  Interventions: Procedure: Surgery
- Surgical group (Active Comparator): In this group, the patients with clinically complete response will undergo surgical treatment (LAR with anal preservation or APR)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgery procedures include LAR+ anal preservation or APR

SUMMARY:
In the present project, the investigators plan to more accurately select the rectal cancer patients with pathological complete response (pCR) to preoperative concomitant chemoradiation therapy (CCRT), taking advantage of quantification of circulating tumor DNA (ctDNA) in addition to the current available diagnostic modalities, including CT, MRI, PET and colonoscopy. The patients with suspected pCR to CCRT will be randomized to radical surgery and local excision groups, followed by the comparison of the oncologic outcomes between two treatment methods. The investigators hypothesized that if the pCR for patients with rectal cancer after CCRT can be more accurately predicted, such patients can be safely treated with limited surgery to enhance the post-treatment life quality, in comparison with patients undergoing radical surgery.

DETAILED DESCRIPTION:
In Taiwan, patients with stage Ⅱ or Ⅲ rectal cancer represented around 30% of all cases of colorectal cancer(n=15,000 annually). Standard treatment of locally advanced rectal cancer consists of neoadjuvant chemoradiotherapy (nCRT), total mesorectal excision (TME), and postoperative adjuvant chemotherapy. This intensive treatment leads to good local tumor control and patient survival, but is associated with short- and long-term morbidity that impairs each patient's quality of life permanently. Although nCRT followed by adjuvant chemotherapy are associated with specific toxicity and may compound surgery-related morbidity, most of the side effects of multimodal treatment that impair the patient's quality of life are attributable to TME with sphincter-preservation or abdomino-perineal resection (APR). Even with the technological advances of robotic and transanal TME, some patients with distal rectal cancer will still require a permanent colostomy. In addition, patients who undergo a sphincter-saving procedure develop a combination of defecatory symptoms known as low anterior resection syndrome. These symptoms are associated with significant impairment of patients' quality of life. With the age-adjusted incidence of rectal cancer increasing steadily in young patients, alternatives to TME are needed.

Some patients with locally advanced rectal cancer have a pathological complete response (pCR) to nCRT. Because patients with pCR have excellent prognosis,8 surgeons question the added value of TME for patients with a clinical complete response (cCR) to CRT. Several institutional case series have reported that a watch-and-wait strategy can result in sustained organ preservation in patients with a cCR to nCRT. Remarkably, up to 30% of patients entered in watch-and-wait protocols eventually experienced tumor re-growth, but most of the cases were surgically salvageable.9 In some series, the survival rate in patients with clinical complete response (cCR) entered in a watch-and-wait protocol was equivalent to that in patients found to have a pCR after TME. However, most of these series, recently published together as an international multicenter registry study, are heterogeneous in terms of tumor stages, radiation dosage, sensitizing chemotherapy, the criteria and timing for assessment of response, and surveillance follow-up protocols. Because these series included only selected patients entering in the watch-and-wait protocol without reporting the total number of patients with similar-stage rectal tumors treated with neoadjuvant therapy during the study period, the possibility of selection bias cannot be excluded. Without a reference denominator, the number of patients who would have potentially benefited from organ preservation by using a watch-and-wait strategy is unknown.

With above-mentioned reasons, most of the patients, including the international case series and our previous case reports, still receive radical surgery for their rectal cancer with cCR to neoadjuvant CRT; some patients with cCR even received a theoretically unnecessary APR procedure and wore a colostoma for life. To enhance the life quality for such patients with cCR to nCRT, the guidelines of the National Comprehensive Cancer Network for treatment of rectal cancer included total neoadjuvant therapy (TNT; systemic chemotherapy before rather than after TME), which was developed in part as a strategy to increase the rate of tumor response. However, to date, the impact of TNT on the potential for organ preservation through avoidance of surgery is unknown.

There is no denying that the organ preservation with no immediate surgery, i.e., the watch-and-wait strategy, in selected patients with a cCR after nCRT is currently at the forefront of rectal cancer management. This strategy is considered as an attractive option to avoid major surgery and the associated morbidity and mortality risks, and functional consequences. However, with the watch-and-wait approach, there is a risk for the development of local regrowth, systemic recurrence, or both, despite the initial achievement of a clinical complete response. Overall, the risk of local re-growth within 3 years from attaining a clinical complete response is 25-30%, and even the occurrence of local re-growth at as long as 7 years from the completion of neoadjuvant chemoradiotherapy has been reported. Therefore, long-term and intensive surveillance protocols have been recommended for patients managed by a watch-and-wait strategy. Remarkably, in consideration of the watch-and-wait policy requires intensive medical resources, it has been not adopted in Taiwan and most of the centers of excellence worldwide.

On the other hand, the GRECCAR2 multicenter randomized trial showed that no evidence of difference in oncological outcomes between local excision and total mesorectal excision in term of 5-year overall survival. Local excision can be proposed in selected patients having a small T2-T3 low rectal cancer with a good clinical response after chemoradiotherapy. However, their study subjects were not limited to rectal cancer with cCR to preoperative CCRT.

The investigators believe that local excision can be applied to the highly selective patients with rectal cancer, especially those with cCR to operative CCRT. However, up to date, there is still no diagnostics to accurately predict the pCR of the rectal cancer to CCRT. And therefore, both the colorectal surgeons and patients has been receiving radical surgery as the major treatment modality. Remarkably, with advent of genetic technology, it become feasible to utilize ctDNA for predicting the response to neoadjuvant chemoradiotherapy and prognosis assessment in locally advanced rectal cancer.

The ctDNA (mutant allele) has been known to be with an extremely short plasma half-life (shorter than 2 hours) compared with tumor markers (such as CEA and CA19-9). After curative resection, therefore, ctDNA rapidly disappears from the blood if no residual cancer exists. Utilizing these characteristics of ctDNA, a diagnostic system for detecting minimal residual disease (MRD) using a next generation sequencing technology is being developed. Remarkably, SignateraTM is a novel ctDNA detection system for MRD detection developed by Natera Inc., U.S.A. First, whole exon analysis of tumor tissue samples is performed, followed by extraction of 16 somatic mutations from the detected tumor-specific single nucleotide variants using an original program, and the primer set that detects these variants is established for each patient and tumor. SignateraTM is a test system that extracts ctDNA from the blood obtained postoperatively, using this primer set, and detects the presence or absence of somatic mutations derived from tumors using a next generation sequencer. In SignateraTM, the sensitivity limit for ctDNA allele frequency is 0.005%, the 90% sensitivity limit is 0.010%, and the specificity is at least 99.5%. In a multicenter prospective cohort study in patients with Stage I-III colorectal carcinoma, 130 patients with Stage I-III colorectal carcinoma were enrolled. The ctDNA positive rate at 30 days after the curative resection was 10.6%, and the relapse rate was 7 times or more higher in the ctDNA positive group than in the ctDNA negative group (hazard ratio [HR] = 7.2; 95% CI, 2.7-19.0). In addition, of the 58 patients who were evaluable for ctDNA after completing postoperative adjuvant chemotherapy, 7 patients (12.0%) were positive for ctDNA, and 51 patients (88.0%) were negative for ctDNA, with relapse observed in all ctDNA-positive patients, which was significantly higher than the relapse rate in ctDNA-negative patients (7/51 patients, 13.7%) (HR = 17.5; 95% CI, 5.4-56.5). Moreover, of the 75 patients who were tested for ctDNA chronologically, 14 out of 15 ctDNA-positive patients (93.3%) had a relapse, and of the 60 patients who were negative for ctDNA, only 2 patients had a relapse. With respect to time-to-relapse, the median time to confirmation of a relapse by ordinary CT scan was 14.2 months, while the median time to detection of positive ctDNA was 5.5 months.

In the present project, the investigators plan to more accurately select the rectal cancer patients with pCR to preoperative CCRT, taking advantage of quantification of ctDNA in addition to the current available diagnostic modalities, including CT, MRI, PET and colonoscopy. The patients with suspected pCR to CCRT will be randomized to radical surgery and local excision groups, followed by the comparison of the oncologic outcomes between two treatment methods. The investigators hypothesized that if the pCR for patients with rectal cancer after CCRT can be more accurately predicted, such patients can be safely treated with limited surgery to enhance the post-treatment life quality, in comparison with patients undergoing radical surgery.

ELIGIBILITY:
Inclusion Criteria:

1. rectal adenocarcinoma completed nCRT and the imaging studies showed no residual malignancy;
2. physical status is within American Society of Anesthesiology（ASA）class Ⅰ to Ⅲ;
3. the lesion side can be reached by the transanal local excision, generally within 6 cm above anal verge;
4. age is 18-75 years.

Exclusion Criteria:

1. Quantification of ct DNA shows residual malignancy;
2. Body mass index（BMI）>40 kg/m2;
3. Previous abdominal or pelvic surgery;
4. abnormal hepatologic (Bil>2.0 mg/dl), renal (Cre≧2.0) and hematologic(WBC<3000, HB<8.0, platelet<50000) profiles after CCRT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-04-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Overall disease-free survival | 3 years
  The duration from surgical resection of primary tumor to the cancer recurrence

SECONDARY OUTCOMES:
Postoperative 30-day complications | 30 days
  Defined as Clavien-Dindo classification. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The class I means no complication, whereas class V means death of the patient.
The length of stay | An average of 7 days
  The duration from the time of surgery to the time of leaving the hospital
Overall survival | 3 years
  The duration from surgical resection of primary tumor to the death due to cancer progression

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung LIANG, MD, Study Director — National Taiwan University Hospital
Locations (1):
- Jin-Tung LIANG, Taipei, Taiwan